CLINICAL TRIAL: NCT00002875
Title: Phase III Prospective Randomized Study of Craniospinal RT Followed by One of Two Adjuvant Chemotherapy Regimens (CCNU, CDDP, VCR OR CPM, CDDP, VCR) for Newly-Diagnosed Average Risk MedulloblastomaMEDULLOBLASTOMA
Brief Title: Radiation Therapy Plus Combination Chemotherapy in Treating Children With Medulloblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Pediatric Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: A9961; CCG-A9961 (Other: Children's Cancer Group); POG-A9961 (Other: Pediatric Oncology Group); CDR0000065160 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Brain Tumors; Central Nervous System Tumors
Keywords: untreated childhood medulloblastoma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cisplatin; Cyclophosphamide; Lomustine; Mesna; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen A (Experimental): Following surgery, craniospinal irradiation followed by a boost to the primary tumor. Beginning within 1 week after initiation of radiotherapy, patients receive vincristine sulfate weekly for 8 doses. Beginning 6 weeks after the completion of radiotherapy, patients receive adjuvant lomustine/vincristine sulfate/cisplatin every 6 weeks for a total of 8 courses.
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: lomustine; Drug: mesna; Drug: vincristine sulfate; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy
- Regimen B (Experimental): Following surgery, craniospinal irradiation plus vincristine sulfate, followed by adjuvant cyclophosphamide/vincristine sulfate/cisplatin every 6 weeks for a total of 8 courses.
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: mesna; Drug: vincristine sulfate; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Biological: filgrastim
  Other Names: G-CSF; Neupogen; NSC-614629
Drug: cisplatin
  Other Names: Platinol; NSC-119875
Drug: cyclophosphamide
  Other Names: Cytoxan; NSC-26271
Drug: lomustine
  Other Names: CCNU; NSC-79037
  Arms: Regimen A
Drug: mesna
  Other Names: Mesnex; NSC-113891
Drug: vincristine sulfate
  Other Names: Oncovin; NSC-67574
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective when combined with radiation therapy for treating medulloblastoma.

PURPOSE: Randomized phase III trial to compare two combination chemotherapy treatments plus radiation therapy in treating children with newly diagnosed medulloblastoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess whether a cyclophosphamide-containing combination chemotherapy regimen increases progression-free survival compared to a lomustine-containing regimen in children with newly diagnosed, average-risk medulloblastoma. II. Determine progression-free and overall survival of children treated with craniospinal radiotherapy and local boost radiotherapy for a total dose of 5580 cGy followed by adjuvant lomustine/cisplatin/vincristine vs. cyclophosphamide/cisplatin/vincristine. III. Determine the long-term neurocognitive, endocrinologic, and cardiopulmonary sequelae associated with craniospinal radiotherapy, local boost radiotherapy, and adjuvant chemotherapy in these children, and determine whether replacement of lomustine with cyclophosphamide alters the incidence and degree of sequelae. IV. Determine whether cellular and biologic parameters, including tumor molecular genetic analysis, DNA ploidy, mitotic activity markers, and immunohistochemical analysis, are correlated with progression-free survival, overall survival, and patterns of disease relapse in these patients. V. Evaluate the utility of routine magnetic resonance imaging surveillance studies of the head and spine in detecting subclinical recurrent disease.

OUTLINE: This is a randomized study. Patients are stratified by participating institution. Following surgery, patients are randomized to one of two groups. The first group receives craniospinal irradiation followed by a boost to the primary tumor. Beginning within 1 week after initiation of radiotherapy, patients receive vincristine weekly for 8 doses. Beginning 6 weeks after the completion of radiotherapy, patients receive adjuvant lomustine/vincristine/cisplatin every 6 weeks for a total of 8 courses. The second group receives craniospinal irradiation plus vincristine as above, followed by adjuvant cyclophosphamide/vincristine/cisplatin every 6 weeks for a total of 8 courses. Patients are followed every 3 months for 1 year, every 6 months for 2 years, then annually.

PROJECTED ACCRUAL: It is anticipated that 240-300 patients will be entered over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Pathologically confirmed posterior fossa medulloblastoma (CCG diagnosis code 2041) Localized disease required, i.e.: No more than 1.5 square centimeters of residual tumor on postoperative contrast-enhanced CT or MRI (preferably within 72 hours but no more than 14 days after surgery) No evidence of metastatic disease on pre- and postoperative MRI of spine (with dye enhancement) and lumbar cerebrospinal fluid (CSF) cytology within 3 days prior to surgery Cytologic analysis of ventricular CSF allowed only if medical contraindication to lumbar puncture and with approval of study chairperson Brain stem involvement eligible

PATIENT CHARACTERISTICS: Age: 3 to 21 at diagnosis Performance status: Not specified Hematopoietic: ANC greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 10 g/dL Hepatic: Bilirubin less than 1.5 mg/dL ALT less than 1.5 times normal Renal: Nuclear glomerular filtration rate or creatinine clearance greater than 70 mL/min per 1.73 square meters

PRIOR CONCURRENT THERAPY: No prior radiotherapy or chemotherapy (other than corticosteroids) No more than 31 days since definitive surgery

Ages: 3 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 421 (Actual)
Dates: Start 1996-12; Primary Completion 2006-02 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Roger J. Packer, MD, Study Chair — Children's National Research Institute; Amar Gajjar, MD, Study Chair — St. Jude Children's Research Hospital
Locations (41):
- United States (36):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Via Christi Regional Medical Center, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico
- Clinique de Pediatrie, Geneva, Switzerland

REFERENCES:
- [Background] Turgut M. Cerebellar mutism. J Neurosurg Pediatr. 2008 Mar;1(3):262. doi: 10.3171/PED/2008/1/3/262. PMID 18352776
- [Background] Robertson PL, Muraszko KM, Holmes EJ, Sposto R, Packer RJ, Gajjar A, Dias MS, Allen JC; Children's Oncology Group. Incidence and severity of postoperative cerebellar mutism syndrome in children with medulloblastoma: a prospective study by the Children's Oncology Group. J Neurosurg. 2006 Dec;105(6 Suppl):444-51. doi: 10.3171/ped.2006.105.6.444. PMID 17184075
- [Result] Packer RJ, Gajjar A, Vezina G, Rorke-Adams L, Burger PC, Robertson PL, Bayer L, LaFond D, Donahue BR, Marymont MH, Muraszko K, Langston J, Sposto R. Phase III study of craniospinal radiation therapy followed by adjuvant chemotherapy for newly diagnosed average-risk medulloblastoma. J Clin Oncol. 2006 Sep 1;24(25):4202-8. doi: 10.1200/JCO.2006.06.4980. PMID 16943538
- [Result] Packer RJ, Gajjar A, Vezina G, et al.: 2340 cGy of craniospinal radiotherapy (CSRT) plus chemotherapy for children with "average-risk" medulloblastoma (MB): a prospective randomized Children's Oncology Group study (A9961). [Abstract] Neuro-Oncology 6 (4): TP-06, 387, 2004.